CLINICAL TRIAL: NCT02987296
Title: A Translational Clinical Trial of Perioperative Immunonutrition in Colorectal Cancer Patients Undergoing Abdominal Surgery: PERIOP-02
Brief Title: Perioperative Immunonutrition in Colorectal Cancer Patients Undergoing Abdominal Surgery
Acronym: PERIOP-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20160732-01H
Record Dates: First submitted 2016-10-25; First posted 2016-12-08 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: ColoRectal Cancer
Keywords: Colorectal Cancer; Surgery; Arginine depletion; Immune system dysfunction; Arginine Supplementation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immunonutrition Diet; Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunonutrition with arginine (Active Comparator): Patients will receive the nutritional supplement for 5 days prior to surgery and for 5 days after. The drink will contain arginine.
  Interventions: Dietary Supplement: Immunonutrition with arginine
- Immunonutrition without arginine (Placebo Comparator): This group of patients will also receive a nutritional drink but containing no arginine for 5 days before surgery and for 5 days after surgery.
  Interventions: Dietary Supplement: Immunonutrition without Arginine

INTERVENTIONS:
Dietary Supplement: Immunonutrition with arginine — Nutritional beverage containing supplemental arginine taken 3 times per day
  Arms: Immunonutrition with arginine
Dietary Supplement: Immunonutrition without Arginine — Nutritional beverage without supplemental arginine taken 3 times per day
  Arms: Immunonutrition without arginine

SUMMARY:
The immune system plays an important role in helping to kill and prevent cancers. Cells of the immune system, such as natural killer (NK) cells and T cells, do not work as well following surgery. Arginine, an amino acid, is fundamental in metabolic processes of the body. Surgery has shown to cause a reduction of arginine in the body. In turn, this deficiency causes NK cell suppression. In this study, we want to look at the effects of arginine supplementation before and after surgery on NK cell function in surgery patients. In this study, we will be using a nutritional supplement containing arginine and a placebo drink (provided by Enhanced Medical Nutrition) that will be taken by colorectal cancer patients 5 days before surgery and 5 days after surgery. Using patient blood samples, we will measure NK cell levels, arginine levels and also arginase activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of a primary colorectal cancer and eligible for surgical resection.
* Patients > 18 years of age
* Eligible patients must have signed a consent for surgical resection of the malignancy.
* Ability to understand and provide a signed informed consent form (ICF) approved by the Research ethics board (REB).
* Adequate kidney function with Creatine clearance>30mL/min
* Hemoglobin level >90 mg/dL
* Ability to comply with protocol requirements.

Exclusion Criteria:

* Prior adjuvant chemotherapy or radiation within 8 weeks of planned surgery.
* Documented significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids, azathioprine, cyclosporin A). Subjects may be on physiologic doses of replacement prednisone or equivalent doses of corticosteroid (<7.5 mg daily).
* Subjects with resting hypotension (Blood pressure <90/50 at rest).
* History of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis.
* Serious intercurrent chronic or acute illness, or other illness considered by the investigator as an unwarranted high risk for an investigational product.
* Active infection of any site and/or active herpes requiring ongoing treatment
* Known pregnancy or nursing mothers
* Subjects with a fish allergy.
* Subjects with severe asthma defined as asthma not controlled with inhaled corticosteroids and additional controllers or by oral corticosteroid treatment (arginine can cause allergic response or make swelling in airways worse).
* Subjects with a known inherited guanidinoacetate methyltransferase deficiency (due to an inability to convert arginine to creatine)
* Subject with known history of liver cirrhosis
* Subjects who have who have suffered a myocardial infarction or life-threatening arrhythmia within the last 6 months
* Subjects with cardiac failure or coronary artery disease causing unstable angina
* Subjects with a medical or psychological impediment to probable compliance with the protocol should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
NK cell killing as measured on peripheral blood mononuclear cells (PBMC) between the control (placebo) and experimental cohorts, using a standard NK cell killing assay. | Baseline (before surgery), post-operative day 1

SECONDARY OUTCOMES:
Decrease in postoperative serum arginine levels between the control (placebo) and experimental cohorts | Baseline (before surgery), post-operative day 1, 3, 5 and 35
Compliance with perioperative arginine supplementation | 5 days preoperatively to 5 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Auer, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Angka L, Martel AB, Ng J, Pecarskie A, Sadiq M, Jeong A, Scaffidi M, Tanese de Souza C, Kennedy MA, Tadros S, Auer RC. A Translational Randomized Trial of Perioperative Arginine Immunonutrition on Natural Killer Cell Function in Colorectal Cancer Surgery Patients. Ann Surg Oncol. 2022 Nov;29(12):7410-7420. doi: 10.1245/s10434-022-12202-y. Epub 2022 Jul 25. PMID 35879482